CLINICAL TRIAL: NCT05269537
Title: Changes in Cardiac Output During Cesarean Delivery Under Spinal Anesthesia. A Prospective Observational Study Using Transthoracic Echocardiography
Brief Title: Changes in Cardiac Output During Cesarean Delivery Under Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Tawfik, Assistant Professor, Department of Anesthesia and Surgical Critical Care, Mansoura University Hospitals, Mansoura, Egypt, Mansoura University
Other Study IDs: MS.20.08.1232
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia, Spinal; Cesarean Section; Echocardiography; Cardiac Output
MeSH Terms: interventions — Anesthesia, Spinal; Cesarean Section; Oxytocin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Cardiac output will be measured at baseline using transthoracic echocardiography. Spinal anesthesia will be administered with injection of intrathecal bupivacaine and intrathecal fentanyl. Crystalloid coload 1000 mL will be administered: Ringer acetate 1000 mL will be administered over 10 minutes starting immediately after intrathecal injection. Cardiac output will be measured at 10 minutes after intrathecal injection, immediately after delivery, at 1 hour after intrathecal injection. Cesarean delivery will be performed. Intravenous ephedrine will be administered to correct hypotension. After delivery, 10 units of oxytocin in 500 ml Ringer acetate will be administered over 30 minutes.
  Interventions: Radiation: Transthoracic Echocardiography; Procedure: Spinal Anesthesia; Drug: Intrathecal Bupivacaine; Drug: Intrathecal Fentanyl; Drug: Crystalloid Coload 1000 mL; Procedure: Cesarean Delivery; Drug: Intravenous Ephedrine; Drug: Oxytocin

INTERVENTIONS:
Radiation: Transthoracic Echocardiography — Measurement of cardiac output in supine position with left lateral tilt at baseline, at 10 minutes after intrathecal injection, immediately after delivery, and at 1 hour after intrathecal injection
Procedure: Spinal Anesthesia — Performed at the L3-L4 or L4-L5 interspace using 25-gauge spinal needle
Drug: Intrathecal Bupivacaine — Bupivacaine 12.5 mg (2.5 mL 0.5%) will be administered in the subarachnoid space
Drug: Intrathecal Fentanyl — Fentanyl 15 μg will be administered in the subarachnoid space
Drug: Crystalloid Coload 1000 mL — Ringer acetate 1000 mL will be administered over 10 minutes starting immediately after intrathecal injection
Procedure: Cesarean Delivery — Lower segment cesarean section using the Pfannenstiel incision and uterine exteriorization
Drug: Intravenous Ephedrine — Intravenous ephedrine 3, 5, and 10 mg will be administered when Systolic blood pressure decreases below 90%, 80%, and 70% of baseline, respectively.
Drug: Oxytocin — Intravenous oxytocin 10 U in 500 mL Ringer acetate will be administered over 30 minutes starting immediately after delivery of the fetus

SUMMARY:
Cardiac output will be measured in healthy parturients undergoing cesarean delivery under spinal anesthesia

DETAILED DESCRIPTION:
ASA-II women undergoing cesarean delivery under spinal anesthesia will be included. Cardiac output will be measured using transthoracic echocardiography at 4 time points: Baseline, after 10 minutes of intrathecal injection, after delivery, and after 1 hour of intrathecal injection. Spinal anesthesia will be administered with 2.5 ml bupivacaine 0.5% and fentanyl 15 μg.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status II parturients.
* Full term, singleton pregnancy
* Elective cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Height <150 cm
* Weight <60 kg
* Body mass index (BMI) <18.5 or ≥ 35 kg/m²
* Women presenting in labor
* Contraindications to spinal anesthesia: increased intracranial pressure, coagulopathy, or local skin infection
* Hemoglobin <10 g/dL
* Current administration of vasoactive drugs (e.g., salbutamol, thyroxin)
* Diabetes mellitus, cardiovascular, or renal disease
* Chronic or pregnancy-induced hypertension
* Polyhydramnios
* Women with high risk for postpartum hemorrhage or uterine atony (e.g., placenta accreta spectrum, ≥3 previous cesarean deliveries)

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy women with full term, singleton pregnancy presenting for elective cesarean delivery under spinal anesthesia in a tertiary obstetric hospital
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
Changes in cardiac output | At baseline, at 10 minutes after intrathecal injection, immediately after delivery, and at 1 hour after intrathecal injection
  Cardiac output measured using transthoracic echocardiography

SECONDARY OUTCOMES:
Changes in stroke volume | At baseline, at 10 minutes after intrathecal injection, immediately after delivery, and at 1 hour after intrathecal injection
Changes in heart rate | At baseline, at 10 minutes after intrathecal injection, immediately after delivery, and at 1 hour after intrathecal injection
Number of subjects requiring ephedrine | From intrathecal injection to the end of cesarean delivery
Incidence of hypotension | From intrathecal injection to the end of cesarean delivery
  Systolic blood pressure <80% of baseline
Incidence of severe hypotension | From intrathecal injection to the end of cesarean delivery
  Systolic blood pressure <70% of baseline
Incidence of bradycardia | From intrathecal injection to the end of cesarean delivery
  Heart rate <50 beats/min
Incidence of nausea and/or vomiting | From intrathecal injection to the end of cesarean delivery
Neonatal Apgar scores | At 1 and 5 minutes after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Tawfik, MD, Principal Investigator — Department of Anesthesia and Surgical Critical Care, Mansoura University Hospitals, Mansoura, Egypt
Locations (1):
- Department of Anesthesia and Surgical Critical Care, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No